CLINICAL TRIAL: NCT05652439
Title: Multinational Database Cohort Study to Assess Adverse Cardiovascular and Cerebrovascular Outcomes in Patients With COPD Initiating a Fixed Triple Therapy Containing BDP, FF and GB Administered Via DPI Compared to pMDI
Brief Title: PASS to Assess Cardiovascular and Cerebrovascular Events in COPD Patients Initiating Fixed Triple Therapy (DPI or pMDI)
Acronym: TRIBE
Status: Recruiting | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-05993BA1-05; EUPAS47420 (Other: EU PAS)
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: retrospective; cardiovascular; cerebrovascular; triple therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fixed triple therapy BDP/FF/GB via DPI: COPD patients new users of fixed triple therapy BDP/FF/GB administered via DPI formulation according to local clinical practice
  Interventions: Other: Observational retrospective data collection
- Fixed triple therapy BDP/FF/GB via pMDI: COPD patients new users of fixed triple therapy BDP/FF/GB administered via pMDI formulation according to local clinical practice
  Interventions: Other: Observational retrospective data collection

INTERVENTIONS:
Other: Observational retrospective data collection — Observational retrospective data collection of the incidence of adverse cardiovascular and cerebrovascular outcomes
  Other Names: No treatment given

SUMMARY:
The aim of this Post Authorisation Safety Study (PASS) is to assess the incidence of adverse cardiovascular and cerebrovascular events in COPD patients who are new to inhaled fixed triple therapy (dual bronchodilator plus corticosteroid) administered via Dry Powder Inhaler (DPI) compared to new users of pressurized Metered Dose Inhaler (pMDI).

Data from clinical practice from different European data sources will be collected. The baseline hypothesis is that the DPI is not associated with different risks of the primary and secondary outcomes, compared with pMDI.

DETAILED DESCRIPTION:
Non-interventional, multi-country cohort study to assess the incidence of adverse cardiovascular and cerebrovascular events among patients with chronic obstructive pulmonary disease (COPD), exposed to inhaled fixed triple therapy BDP/FF/GB via DPI (drug of interest) or pMDI (comparator).

The study will be conducted based on secondary health data collected (as per clinical practice) retrospectively from seven different European data sources in the following countries: United Kingdom, Germany, The Netherlands, Denmark, Sweden, Norway and Finland.

Patients in the two exposure groups of this Post Authorisation Safety Study (PASS) will be followed for the study outcomes from the start of the exposure until the first occurrence of end of treatment, switch to the other study drug, end of the study period, or censoring. The pre-defined hypothesis is that the DPI is not associated with different risks of the primary and secondary outcomes, compared with pMDI.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD
* 40 years or older
* Availability of baseline information for a minimum of 12 months before the index date
* New users of single inhaler triple therapy BDP/FF/GB via DPI or pMDI

Exclusion Criteria:

* Single or multi-inhaler triple therapy in the previous 90 days before the index date
* Prescription of BDP/FF/GP administered via pMDI or DPI or any other single inhaler triple therapy in addition to a study drug on the index date.
* Hospitalization due to cardiovascular causes in the previous 30 days before the index date.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients diagnosed with COPD, aged 40 years or older. Eligible for inclusion will be patients with new use of single inhaler triple therapy BDP/FF/GB via DPI or pMDI and no use of any single or multi-inhaler triple therapy (including the study drugs) in the previous 90 days.
  The source population includes patients who have at least one prescription/dispensation of BDP/FF/GB administered via DPI or pMDI during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | Through study completion, up to 5 years
  To assess the incidence of MACEs and compare it between fixed triple therapy BDP/FF/GB via DPI and pMDI formulation. MACEs will be defined as any of the following events:
  * Myocardial infarction
  * Stroke (ischemic and haemorrhagic stroke)
  * Hospitalization due to acute coronary syndrome
  * Hospitalization due to heart failure

SECONDARY OUTCOMES:
Incidence of major cardiovascular and cerebrovascular events individually | Through study completion, up to 5 years
  To assess the incidence of each of the following events individually:
  * Myocardial infarction
  * Cerebrovascular disorders (ischemic and haemorrhagic stroke, transient ischemic attack)
  * Hospitalization due to acute coronary syndrome
  * Hospitalization due to heart failure
  * Arrhythmias (new-sustained supra-ventricular and sustained ventricular)
  * All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Hoti, Principal Investigator — Iqvia Pty Ltd
Locations (1):
- Clinical Practice Research Datalink (CPRD), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be analysed in this study